CLINICAL TRIAL: NCT04104854
Title: Safety and Efficacy of Drug Coated Balloon Therapy for de Novo Lesions in Patients With Coronary Heart Disease Under the Guidance of QFR (UNIQUE-DCB-I Study )
Brief Title: Safety and Efficacy of DCB Therapy for de Novo Lesions Under the Guidance of QFR in CHD Patients (UNIQUE-DCB-I Study )
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY201909
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Coronary Heart Disease
Keywords: Quantitative flow ratio; drug coated balloon; Drug eluted stent; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- drug coated balloon (Experimental): A total of 110 patients are assigned to drug coated balloon treated group after randomization schedule.
  Interventions: Device: drug coated balloon
- drug eluted stent implantation (No Intervention): A total of 110 patients are assigned to drug eluted stent treated group after randomization schedule.

INTERVENTIONS:
Device: drug coated balloon — Balloon/vessel diameter ratio 0.8-1.0, 8-12 ATM (atmosphere), lasting for >30 seconds
  Arms: drug coated balloon

SUMMARY:
Since Gruntzig successfully performed percutaneous coronary balloon angioplasty in 1977, percutaneous coronary intervention has developed rapidly. From bare metal stents to drug-eluting stents (DES), the symptoms and prognosis of patients with coronary heart disease (CHD) have been greatly improved. Although DES has reduced the probability of in-stent restenosis (ISR) and thrombosis compared with BMS since its clinical application, it can not completely solve this problem. Even if the new generation of DES requires revascularization, the incidence of ISR is still as high as 5%-10%. DES treatment is associated with delayed endothelial healing, late acquired poor stent adherence and new atherosclerosis, which lead to late ISR and thrombosis. In addition, DES is still not ideal for the treatment of small vessel disease, diffuse long lesion and bifurcation lesion. Therefore, drug coated balloon (DCB) has attracted people's attention. Balloon-loaded antiproliferative drugs can fully release the drugs to the vascular wall during balloon dilation, which can inhibit the restenosis process from the beginning of injury, and show good efficacy and safety in some specific lesions. Many clinical studies have shown that DCB has good efficacy and safety in some specific lesions (ISR, small vessel disease, bifurcation disease, in situ lesion). Especially in the treatment of ISR, researchers believe that its efficacy is not inferior to DES, and it has the advantage of non-metal residues.

Quantitative flow ratio (QFR) is the second generation FFR detection method based on angiographic images. The diagnostic accuracy of QFR 0.80 for myocardial ischemic stenosis was 92.7%. Compared with QCA, the positive predictive value and negative predictive value of QFR were also significantly better than those of QCA. The latest FAVOR II results also confirm that QFR is more sensitive and specific in diagnosing myocardial ischemia caused by coronary artery stenosis than QCA, and confirm the feasibility of using QFR online in catheter lab to evaluate the functional significance of coronary artery critical lesions. However, there is no report on the treatment of de novo lesions in patients with coronary heart disease by DCB under the guidance of QFR. The aim of this study was to evaluate the safety and efficacy of drug balloon therapy for de novo lesions in patients with CHD under the guidance of QFR compared with DES implantation.

DETAILED DESCRIPTION:
The current study is designed as a multicenter, randomized and prospective study aiming to evaluate the safety and efficacy of drug balloon therapy for de novo lesions in patients with CHD under the guidance of QFR compared with DES implantation. Based on previous study, the incidence rate of target lesion failure is 5%-10% in patients with CHD undergoing DES implantation. And in the investigators study the expected incidence rate of target lesion failure is up to 5.0 % in patients with CHD after treatment with DCB. Moreover, the investigators estimated 10% loss follow-up of these patients in each arm. As a result, a total of 220 patients with CHD were required, and with 110 patients per group as a ratio of 1:1 randomization.

ELIGIBILITY:
Inclusion Criteria:

●Meet the diagnostic criteria for stable angina pectoris, unstable angina pectoris and acute myocardial infarction and QFR<0.8 of target lesion

Exclusion Criteria:

* QFR less than 0.8, dissection above type B and thrombosis formation after pre-dilation of coronary artery lesions
* Severe congestive heart failure [LVEF <30% or NYHA( New York Heart Association) III/IV)]
* Severe valvular heart disease
* Life expectancy no more than 1 year or factors causing difficulties in clinical follow up
* Intolerance to aspirin and/or clopidogrel
* Known intolerance or allergy to heparin, contrast agents, paclitaxel, iopromide, rapamycin, polylactic acid-glycolic acid copolymer, Co-Cr alloy or platinum-chromium alloy
* Leukopenia or thrombopenia
* A history of peptic ulcer or GI bleeding in the previously
* Stroke within 6 months prior to the operation
* A history of severe hepatic or renal failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of late lumen loss after percutaneous coronary intervention in patients with CHD | Follow-up coronary angiography at 12 months after the procedure
  The incidence rate of late lumen loss between DCB treated group and DES treated group evaluated by quantitative coronary analysis in patients with CHD

SECONDARY OUTCOMES:
The incidence rate of device-related ischemic events | Clinical follow up at 30 days, 6, 9 and 12 months after the procedure
  The incidence rate of device-related ischemic events including cardiovascular death, target vessel related myocardial infarction and ischemia-driven revascularization between DCB treated group and DES treated group
The incidence rate of patient-related ischemic events | Clinical follow up at 30 days, 6, 9 and 12 months after the operation
  The incidence rate of patient-related ischemic events including all myocardial infarction , any revascularization and all-cause death between DCB treated group and DES treated group

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ye, MD, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Background] de la Torre Hernandez JM, Garcia Camarero T, Lozano Ruiz-Poveda F, Urbano-Carrillo CA, Sanchez Perez I, Cano-Garcia M, Saez R, Andres Morist A, Molina E, Pinar E, Torres A, Lezcano EJ, Gutierrez H, Arnold RJ, Zueco J. Angiography and Optical Coherence Tomography Assessment of the Drug-Coated Balloon ESSENTIAL for the Treatment of In-Stent Restenosis. Cardiovasc Revasc Med. 2020 Apr;21(4):508-513. doi: 10.1016/j.carrev.2019.07.021. Epub 2019 Jul 23. PMID 31401071
- [Background] Rissanen TT, Uskela S, Eranen J, Mantyla P, Olli A, Romppanen H, Siljander A, Pietila M, Minkkinen MJ, Tervo J, Karkkainen JM; DEBUT trial investigators. Drug-coated balloon for treatment of de-novo coronary artery lesions in patients with high bleeding risk (DEBUT): a single-blind, randomised, non-inferiority trial. Lancet. 2019 Jul 20;394(10194):230-239. doi: 10.1016/S0140-6736(19)31126-2. Epub 2019 Jun 13. PMID 31204115
- [Background] Bech GJ, Pijls NH, De Bruyne B, Peels KH, Michels HR, Bonnier HJ, Koolen JJ. Usefulness of fractional flow reserve to predict clinical outcome after balloon angioplasty. Circulation. 1999 Feb 23;99(7):883-8. doi: 10.1161/01.cir.99.7.883. PMID 10027810
- [Background] Xu B, Tu S, Qiao S, Qu X, Chen Y, Yang J, Guo L, Sun Z, Li Z, Tian F, Fang W, Chen J, Li W, Guan C, Holm NR, Wijns W, Hu S. Diagnostic Accuracy of Angiography-Based Quantitative Flow Ratio Measurements for Online Assessment of Coronary Stenosis. J Am Coll Cardiol. 2017 Dec 26;70(25):3077-3087. doi: 10.1016/j.jacc.2017.10.035. Epub 2017 Oct 31. PMID 29101020